CLINICAL TRIAL: NCT03777020
Title: Evaluating the Efficacy of a Service Dog Training Program for Military Veterans With PTSD
Brief Title: Service Dog Training Program for Military Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Erika Friedmann, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00083872
Record Dates: First submitted 2018-12-10; First posted 2018-12-17 (Actual); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-02

CONDITIONS: Post Traumatic Stress Disorder
Keywords: human-animal interaction; service dog; stress
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Human-Animal Interaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Service Dog Training Program (SDTP) (Experimental): Veterans randomized to the SDTP will be paired with an experienced Warrior Canine Connection (WCC) Mission Based Trauma Recovery (MBTR)-Trainer (MBRT-T) and a service dog (SD). One hour training modules will be scheduled once a week for 8 weeks. Participants will come to WCC for all the weekly training modules. Participants will be paired with the same SD for the duration of the SDTP unless an unforeseen circumstance arises and the SD needs to be removed from the SDTP. The MBTR-T will deliver the prescribed SDTP modules created by WCC. Each session will be fully supervised by a WCC MBTR-T to address any concerns or safety issues that may arise.
  Interventions: Behavioral: Service Dog Training Program
- Dog Training Education (Other): Veterans randomized to Dog Training Education will participate in one hour online SD training modules (https://e-trainingfordogs.com) scheduled once a week for 8 weeks. The online training modules are delivered by experienced SD trainers and will employ parallel content to the WCC SDTP. Participants will come to the WCC site for all the weekly online training modules. Members of the WLCI group will have education about dog training, but NO interaction with a SD. The online training modules for the DTE group are intended to keep the veterans who are not immediately assigned to the SDTP engaged in the study. They will participate in the SDTP after conclusion of participation in the 8 week study.
  Interventions: Other: Dog Training Education

INTERVENTIONS:
Behavioral: Service Dog Training Program — Participate in 8 weekly dog training sessions using a positive reinforcement method and curriculum under the direct supervision of trainer at the Warrior Canine Connection facility in Boyds (Montgomery County) MD.
  Arms: Service Dog Training Program (SDTP)
Other: Dog Training Education — Learn about training dogs by watching 8 weekly dog training online modules programs at the Warrior Canine Connection facility in Boyds (Montgomery County) MD. After completing this education the participants will participate in the service dog training program.
  Arms: Dog Training Education

SUMMARY:
Post-traumatic stress disorder (PTSD), an invisible wound of war, affects approximately 20%1 of the 18.5 million U.S. veterans and places them at higher risk for impaired biopsychosocial functioning. PTSD symptom severity (PTSDSS) is significantly correlated with stress and psychosocial consequences of inability to regulate emotions, control impulsive behaviors, and function within family and society. Alarming veteran PTSD rates and its insidious effects demand empirically validated treatment programs. More than a million veterans receive new diagnoses of each year. VA PTSD therapy programs reach only 1% of veterans. Nearly 35% of veterans do not respond to widely used psychotherapy and pharmacotherapy treatments. Training a service dog (SD) is a novel rehabilitative animal-assisted intervention that shows promise in other populations. This project evaluates the efficacy of a service dog training program (SDTP) as an alternative and adjunctive treatment and rehabilitative option for veterans with PTSD.

DETAILED DESCRIPTION:
Veterans with PTSD attend 8 weekly sessions of either training a service dog or learning about how to train a dog at the Warrior Canine Connection facility in Boyds MD. They complete questionnaires prior to the start of the program and at the midpoint (after 4 sessions) and end of the program (after 8 sessions). Participants also wear a monitor to record heart rate variability during the 1st, 4th, and 8th sessions and provide saliva samples at these same times.

ELIGIBILITY:
Inclusion Criteria

1. Accepted into the Warrior Canine Connection Service Dog Training Program. Their inclusion criteria are:

   1. military veteran;
   2. diagnosis of PTSD;
   3. able to give informed consent; and
   4. able to understand English; And
2. Military Veteran

Exclusion Criteria:

Excluded from the Warrior Canine Connection Service Dog Training Program. Their criteria are:

1. fear of dogs;
2. allergy to pet dander;
3. active substance abuse;
4. active psychosis, or
5. history of animal abuse
6. Excluded by the WCC from participation in their Service Dog Training Program because they have:

fear of dogs; allergy to pet dander; active substance abuse; active psychosis, history of animal abuse or physically unable to complete tasks required to train dogs

.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erika Friedmann, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Warrior Canine Connections, Boyds, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Service Dog Training Program (SDTP) | Dog Training Education
Started | 30 | 30
Completed | 26 | 25
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 4 | 4
Not completed — No longer met inclusion criteria at initial visit | 0 | 1

BASELINE CHARACTERISTICS:
Population: One participant in the dog training education group no longer met inclusion criteria at first visit and was removed from the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Service Dog Training Program (SDTP) | Dog Training Education | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 26 | 54
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (10.5) | 47.3 (12.4) | 47.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 17 | 14 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 30 | 26 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 20 | 19 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Post Traumatic Stress Symptom Severity
Description: Post traumatic stress disorder checklist for DSM-5 range of scores 0-80; higher score is worse (more PTSD)
Time Frame: Baseline, 8 weeks
Population: Veterans with PTSD
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Service Dog Training Program (SDTP) | Dog Training Education
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline: number analyzed (Participants) | 30 | 29
  Baseline | 43.7 (3.1) | 38.9 (3.2)
  8 weeks: number analyzed (Participants) | 26 | 25
  8 weeks | 35.1 (3.1) | 31.6 (3.2)

2. Secondary Outcome: Stress Biomarker Markers:Cortisol
Description: salivary cortisol ug/dL; higher is more stress
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Stress Biomarkers: Alpha Amylase
Description: salivary alpha amylase U/mL; higher is more stress
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Stress Biomarkers: IgA
Description: salivary immunoglobulin A μg/mL; higher is less stress
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Stress Biomarkers: HRV
Description: Heart rate variability Polar H7 heart rate sensor worn around the chest and matching Polar V800 GPS Sports Watch, higher is better
Time Frame: baseline, 8 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Stress Marker: Perceived Stress
Description: Patient Reported Outcomes Measurement Information System (PROMIS) Perceived Stress; PROMIS PS, score range 10 to 50, T scores range from 22.7 to 87.1, higher is more stress perceived
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Psychosocial Health: Positive Affect
Description: PROMIS Positive Affect Short Form 15 (PA 152), raw scores range from 15 to 75 they are converted to T scores range of 14.4 to 69.9 with a mean of 50 and SD or 10, higher is greater positive affect
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Psychosocial Health: Health Related Quality of Life
Description: Veterans RAND 12 Item Health Survey (VR-12); physical health and mental health subscales; scales are calculated with an algorithm with a mean of 50 as the 50th percentile of the U.S. population; higher score is better (higher quality of life).
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Psychosocial Health: Resilience
Description: Connor-Davidson Resilience Scale (CD-RISC-10), scores range from 0 to 40, higher score is more resilient
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Psychosocial Health: Relationship With Friends and Family
Description: Relationship Scale Questionnaire (RSQ) , 4 subscales are created from average of items: Secure scale is the average of 3, 9(Reverse),10, 15, 28(Reverse). Fearful scale is the average of 1, 5, 12, 24. Preoccupied scale is the average of 6(Reverse), 8, 16, 25. Dismissing scale is the average of 2, 6, 19, 22, 26. Subscale scores range from 1 to 5. Higher scores are poorer relationships
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Psychosocial Health: Quality of Individual's Relationships
Description: PROMIS Satisfaction with Social Roles and Activities (SSRA)-Short Form 4a (PROMIS-SSRA), raw scores range from 4 to 20, T scores range from 27.9 to 63.8, higher score is more satisfaction
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Psychosocial Health: Satisfaction With Social Activities
Description: PROMIS Short Form v1.0- Satisfaction with Participation in Discretionary Social Activities- Short Form 7a (PROMIS SPDSA) raw scores range from 7 to 35, T scores range from 28.7 to 67.3, higher score is more satisfaction
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Psychosocial Health: Companionship
Description: PROMIS Companionship - Short Form 4a (PROMIS-C) raw scores range from 4 to 20, T scores range from 25.2 to 65.3, higher score is more companionship
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Psychosocial Health:Depression
Description: PROMIS Depression Short-Form 8a (PROMIS-D), raw scores range from 8 to 40, T scores range from 0-100, higher score is more depression
Time Frame: baseline, 8 weeks
Reporting Status: Not Posted

15. Secondary Outcome: Psychosocial Health: Anxiety
Description: PROMIS Anxiety Short-Form 8a (PROMIS-A) raw scores range from 8 to 40, T scores range from 0-100, higher score is more anxiety
Time Frame: baseline, 8 weeks
Reporting Status: Not Posted

16. Secondary Outcome: Psychosocial Health: Suicidal Ideation
Description: Beck Scale for Suicide Ideation (BSSI), raw scores range from 0 to 38, higher score is greater suicidal ideation
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Cellular Aging
Description: total telomere length (kilobase pairs, from saliva sample) longer telomere length is less cellular aging
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Service Dog Training Program (SDTP) | Dog Training Education
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT03777020/Prot_SAP_000.pdf